CLINICAL TRIAL: NCT07261215
Title: A Study on the Efficacy and Safety of Zuberitamab as First-Line Preemptive Therapy for EBV Infection Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Zuberitamab for EBV Infection Post-Allo-HSCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025118
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: HSCT; EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zuberitamab treatment (Experimental)
  Interventions: Drug: Zuberitamab

INTERVENTIONS:
Drug: Zuberitamab — Zuberitamab will be administered as first-line preemptive therapy at a dose of 375 mg/m² on day 1 of each cycle (one cycle = 7 days).

SUMMARY:
EBV DNAemia is defined as the presence of EBV-DNA load in peripheral blood exceeding the normal threshold, serving as a key diagnostic indicator for EBV-associated post-transplant lymphoproliferative disorder (EBV-PTLD). According to the European Conference on Infections in Leukemia (ECIL-6) guidelines, regular monitoring of peripheral blood EBV-DNA levels via quantitative real-time PCR (qPCR) is recommended starting from the first month after allogeneic hematopoietic stem cell transplantation (allo-HSCT), with a weekly frequency sustained for at least 4 months post-transplant. For HSCT patients who develop EBV DNAemia, preemptive therapy should be initiated promptly. EBV-PTLD is a serious complication that may progress rapidly; if not diagnosed and treated in a timely manner, mortality rates can reach 60-80%. Current guidelines recommend CD20 monoclonal antibody (rituximab) as the first-line preemptive treatment. The response rate to rituximab is approximately 84%. The typical regimen consists of 375 mg/m² per dose, administered weekly, with 1-4 doses generally sufficient to achieve treatment goals. However, a subset of patients exhibits poor response to first-line therapy and requires second-line interventions, such as EBV-specific cytotoxic T lymphocytes (EBV-CTLs), donor lymphocyte infusion, or combination chemotherapy.

Zuberitamab is a novel anti-CD20 monoclonal antibody and the first Class 1 innovative biologics targeting CD20 developed in China. Preclinical studies have demonstrated that zuberitamab exhibits stronger antibody-dependent cellular cytotoxicity (ADCC) activity compared to rituximab. In a pivotal Phase III registrational clinical study, zuberitamab combined with CHOP (Hi-CHOP) was evaluated head-to-head against R-CHOP in patients with diffuse large B-cell lymphoma (DLBCL). The results showed an improvement in the complete response (CR) rate by more than 8% (85.7% vs. 77.3%, P = 0.038). These findings indicate that zuberitamab holds significant advantages over rituximab in terms of both biological activity and clinical efficacy. Based on this evidence, we have initiated a Phase II clinical trial to evaluate the efficacy and safety of zuberitamab as first-line preemptive therapy for EBV infection. This is a prospective Phase II clinical trial enrolling patients with EBV infection following transplantation. Zuberitamab will be administered as first-line preemptive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent allogeneic hematopoietic stem cell transplantation (HSCT).
2. Documented EBV infection, defined as either:

   EBV DNAemia (EBV-DNA ≥400 copies/mL in plasma), or Pathologically confirmed EBV-associated lymphoproliferative disease with positive EBER by in situ hybridization.
3. Age ≥18 years, regardless of gender.
4. Negative for HIV, HBV, and HCV.
5. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0-2.
6. Provision of signed informed consent prior to any study-related procedures. For patients aged 18 or above, consent must be provided by the patient themselves or an immediate family member. If obtaining consent directly from the patient is deemed medically detrimental to their condition, consent may be provided by a legal guardian or an immediate family member.

Exclusion Criteria:

* 1. Presence of uncontrolled infection requiring mechanical ventilation or hemodynamic instability at the time of enrollment.

  2. Diagnosis of clinically significant severe hepatic insufficiency (defined as Child-Pugh Class C) within 5 days prior to enrollment.

  3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding 5 times the upper limit of normal (ULN), or serum total bilirubin exceeding 2 times ULN, within 5 days prior to enrollment.

  4. Diagnosis of end-stage renal dysfunction with a creatinine clearance rate of <10 mL/min within 5 days prior to enrollment.

  5. Concurrent diagnosis of moderate hepatic insufficiency (defined as Child-Pugh Class B) and moderate renal dysfunction (defined as creatinine clearance rate <50 mL/min).

  6. Cardiac function or disease meeting any of the following criteria:
  1. Long QT syndrome or QTc interval >480 ms.
  2. Complete left bundle branch block, second-degree or third-degree atrioventricular block.
  3. Severe, uncontrolled arrhythmia requiring pharmacological intervention.
  4. New York Heart Association (NYHA) functional classification ≥ Class II.
  5. Left ventricular ejection fraction (LVEF) <50%.
  6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia, or any other clinically significant arrhythmia requiring treatment within 6 months prior to enrollment; history of clinically significant pericardial disease; or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

     7. Presence of uncontrolled severe acute graft-versus-host disease (aGVHD). 8. Evidence of active HIV replication prior to enrollment; detectable HCV antibody and HCV-RNA positivity within 90 days prior to enrollment; or HBsAg positivity. Known seropositivity for HIV or active hepatitis C virus.

     9. Presence of psychiatric disorders or other conditions that would compromise the patient's ability to comply with study treatment and monitoring requirements.

     10. Inability or unwillingness to provide written informed consent. 11. Patients deemed ineligible by the investigator due to other specific circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA clearance rate | 28 days after treatment

SECONDARY OUTCOMES:
overall survival (OS) | 180days
relapse-free survival (RFS) | 180 days
Treatment-related mortality | 180 days
Incidence of post-transplant lymphoproliferative disease (PTLD) | 180 days
Incidence of hemophagocytic syndrome | 180 days
Infection rates | 180 days
use of second-line therapy of anti-EBV | 180 days
AE | 180 days
  incidence of adverse events as assessed by the NCI CTCAE version 5.0 criteria